CLINICAL TRIAL: NCT05404412
Title: The Impact of Contrast Media Used In Epidural Steroid Injections on Thyroid Function Tests
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 07.01.2022.83
Record Dates: First submitted 2022-05-29; First posted 2022-06-03 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Lumbar Radiculopathy; Lumbar Spinal Stenosis; Cervical Radiculopathy; Cervical Stenosis
Keywords: thyroid functions; epidural steroid injections
MeSH Terms: conditions — Radiculopathy; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Epidural Steroid Injection — This intervention is applied mostly for cervical or lumbar radiculopathy. The intervention was carried out under sterile conditions with the C-arm fluoroscopy guidance. It is performed via spinal needle and the needle is inserted into the epidural space, then a combined local anesthetic and glucocorticoids are delivered to the epidural space.

SUMMARY:
This study is aim to disclose the effect of contrast media, which used in epidural steroid injections, on the parameters of thyroid function tests (TFTs). The patients who underwent an epidural steroid injection were included. The investigators hypothesized that contrast media owing to contain iodine may impair the values of TFTs.

DETAILED DESCRIPTION:
The objective of this study is to reveal the impact of contrast media, whether they change the values of TFTs in participants who had been performed any kind of epidural steroid injection such as Lumbar, cervical and caudal epidural steroid injection. The inclusion criteria were participants who had normal values of TFTs, being between the ages of 18 and 65 and had an epidural steroid injection. Patients with impaired parameters of TFTs or had thyroid surgery, systemic and/or local infections, malignancy, bleeding diathesis, acute fracture, known allergy to contrast material and/or local anesthetic substances, known history of any psychiatric disorder, and patients with a history of pregnancy were excluded from the study. Verbal and written informed consent was obtained from all patients participating in the study.

In conjunction with the recording of the demographic data of the patients participating in this study (age, sex, duration of symptoms, etc.), their contrast medium doses and the values of TFTs (free T3, free T4 and Thyroid-stimulating hormone) were employed before the procedure and 3rd week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be performing with an epidural steroid injection
* Being between the ages of 18 and 65
* Having normal values of Thyroid function tests

Exclusion Criteria:

* Patients with a history of thyroid surgery or impaired thyroid function tests
* Patients with systemic and/or local infections,
* Malignancy,
* Bleeding diathesis,
* Acute fracture,
* Known allergy to contrast material and/or local anesthetic substances,
* Known history of any psychiatric disorder
* Patients with a history of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, between the ages of 18 and 65, who have normal values of thyroid function tests and who will be performing an epidural steroid injection.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
The Values of free T4 | Change of the values of free T4 from baseline to each checkpoints from pre-interventional time to postinterventional 3rd week
  Free T4 is a type of thyroid hormone. A free T4 test is used to evaluate thyroid function
The Values of free T3 | Change of the values of free T3 from baseline to each checkpoints from pre-interventional time to postinterventional 3rd week
  The free T3 is an another major hormone of the thyroid gland. It is used to show thyroid functions.
The Values of Thyroid-stimülating hormone (TSH) | Change of the values of TSH from baseline to each checkpoints from pre-interventional time to postinterventional 3rd week
  TSH is secreted from the pituitary gland to stimulate the thyroid gland. It regulates thyroid functions. This test is also used for thyroid functions.

CONTACTS AND LOCATIONS:
Overall Officials: SAVAS SENCAN, Principal Investigator — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Knezevic NN, Navani A, Christo PJ, Limerick G, Calodney AK, Grider J, Harned ME, Cintron L, Gharibo CG, Shah S, Nampiaparampil DE, Candido KD, Soin A, Kaye AD, Kosanovic R, Magee TR, Beall DP, Atluri S, Gupta M, Helm Ii S, Wargo BW, Diwan S, Aydin SM, Boswell MV, Haney BW, Albers SL, Latchaw R, Abd-Elsayed A, Conn A, Hansen H, Simopoulos TT, Swicegood JR, Bryce DA, Singh V, Abdi S, Bakshi S, Buenaventura RM, Cabaret JA, Jameson J, Jha S, Kaye AM, Pasupuleti R, Rajput K, Sanapati MR, Sehgal N, Trescot AM, Racz GB, Gupta S, Sharma ML, Grami V, Parr AT, Knezevic E, Datta S, Patel KG, Tracy DH, Cordner HJ, Snook LT, Benyamin RM, Hirsch JA. Epidural Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Comprehensive Evidence-Based Guidelines. Pain Physician. 2021 Jan;24(S1):S27-S208. PMID 33492918
- [Background] Kim YU, Kim D, Park JY, Choi JH, Kim JH, Bae HY, Joo EY, Suh JH. Method to Reduce the False-Positive Rate of Loss of Resistance in the Cervical Epidural Region. Pain Res Manag. 2016;2016:9894054. doi: 10.1155/2016/9894054. Epub 2016 Mar 29. PMID 27445637
- [Background] Kornelius E, Chiou JY, Yang YS, Peng CH, Lai YR, Huang CN. Iodinated Contrast Media Increased the Risk of Thyroid Dysfunction: A 6-Year Retrospective Cohort Study. J Clin Endocrinol Metab. 2015 Sep;100(9):3372-9. doi: 10.1210/JC.2015-2329. Epub 2015 Jul 13. PMID 26168278